CLINICAL TRIAL: NCT06488690
Title: Effectiveness of Early Warning Scores: Preoperative Period in Pregnant Women
Brief Title: Early Warning Scores in Pregnant Woman
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Onurcan BALIK, Doctor, Suleyman Demirel University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: SuleymanDU-MD-OB-01
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Complications
Keywords: Early Warning Scores; MEOWS; MEWC; MEWT; Pregnant Women; Maternal Morbidity
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: Pregnant woman
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients who are pregnant and undergo cesarean section (Other): We included all patients who were pregnant and underwent cesarean section and calculated maternal early warning scores.
  Interventions: Other: All patients who were pregnant and underwent cesarean section

INTERVENTIONS:
Other: All patients who were pregnant and underwent cesarean section — Our study aims to evaluate the use of early warning scores as a screening tool to predict obstetric mortality and morbidity in pregnant women who will undergo cesarean section.

SUMMARY:
Our study aims to evaluate the use of early warning scores as a screening tool to predict obstetric mortality and morbidity in pregnant women who will undergo cesarean section.

DETAILED DESCRIPTION:
Our study aims to evaluate the use of early warning scores as a screening tool to predict obstetric mortality and morbidity in pregnant women who will undergo cesarean section.

This prospective study included 304 patients undergoing cesarean section at Suleyman Demirel University between April 2022 and April 2023. Physiological parameters were assessed in all 304 pregnant women before the operation. Maternal early warning scores, including modified early obstetric warning score (MEOWS), maternal early warning score (MEWC), and maternal early warning triggers (MEWT), were calculated for each patient. Patients triggering the system were classified as Group 1 (risky patients), while those not triggering the system were classified as Group 2 (risk-free patients).

ELIGIBILITY:
Inclusion Criteria:

* All patients who are pregnant and undergo cesarean section

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant Woman
Enrollment: 304 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
MEOWS, MEWC and MEWT scores | One year
  The presence of a "trigger" for MEOWS in all systems, defined as either a single severely abnormal parameter (falling in the "red" zone) or two slightly abnormal parameters (falling in the "yellow" zone), was categorized as the risky group. Absence or mildness of the trigger was considered as the risk-free group.
MEWC score | One year
  In the case of MEWC, the presence of only one abnormal parameter designated the risk group, while the absence of a trigger indicated the risk-free group.
MEWT score | One year
  For MEWT, the presence of a "trigger" defined as either a single severely abnormal parameter (falling in the "red" zone) or two mildly abnormal parameters (falling in the "yellow" zone) was categorized as the risky group, with the absence or mildness of the trigger considered as the risk-free group.

SECONDARY OUTCOMES:
APGAR score | One year
  APGAR scores at 1st and 5th minutes were calculated for postnatal babies.
Aldrete score | One year
  The Modified Aldrete Recovery Score System was computed for mothers to assess postoperative recovery.
Glasgow Coma Scale | One year
  The Glasgow Coma Scale (GCS) was used to evaluate the consciousness of pregnant women.

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University, Isparta, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No